CLINICAL TRIAL: NCT01529385
Title: Efficacy of a Mild Compression Diabetic Sock Versus A Non- Compression Diabetic Sock in the Control of Lower Extremity Edema in Patients With Diabetes: A Randomized Controlled Trial
Brief Title: Mild Compression Sock for Control of Lower Extremity Edema in Individuals With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rosalind Franklin University of Medicine and Science (Other)
Collaborators: Madigan Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dr. Stephanie Wu, DPM, MS, Director of Center for Lower Extremity Ambulatory Research, Rosalind Franklin University of Medicine and Science
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: ORT 112
Record Dates: First submitted 2012-02-03; First posted 2012-02-08 (Estimated); Results first posted 2016-06-22 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-05

CONDITIONS: Edema
Keywords: swollen leg; diabetes; compression stockings; edema
MeSH Terms: conditions — Edema; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mild Compression Diabetic Sock (Experimental): Diabetic socks that provide 18-25mm Hg of pressure to the lower extremities.
  Interventions: Device: mild compression diabetic sock
- Standard Diabetic Sock (Other): A standard diabetic sock that is designed to limit foot ulcer formation, but does not provide compression to the leg.
  Interventions: Device: Standard diabetic sock

INTERVENTIONS:
Device: mild compression diabetic sock — A diabetic sock that provides mild compression (18-25mm Hg) is to be worn everyday for four weeks
  Arms: Mild Compression Diabetic Sock
Device: Standard diabetic sock — A diabetic sock that is not designed to provide compression is to be worn everyday for four weeks
  Arms: Standard Diabetic Sock

SUMMARY:
The purpose of this study is to determine whether a specially designed sock for people with diabetes and swelling in the legs can reduce the swelling, improve blood flow to the legs, and improve physical activity patterns of those individuals by providing mild compression to their legs.

DETAILED DESCRIPTION:
Peripheral arterial disease (PAD) is commonly associated with diabetes. Clinicians are often reluctant to apply compressive stockings to patients with diabetes and swollen legs due to fear of exacerbating the symptoms of PAD. The study sock is a newly formulated sock that offers mild compression (18-25mmHg). The sock is made especially for the diabetic patient who suffers from concomitant lower extremity edema.

Eighty patients with diabetes and lower extremity edema will be recruited. Upon ensuring enrollment criteria are met, baseline edema (as measured by circumference of foot, ankle and calf), ankle brachial index (ABI), skin perfusion pressure, and cutaneous fluid level (as measured by MoistureMeter) will be assessed. Subjects will then be provided four pairs of socks. Subjects will be randomized in a 1:1 distribution to receive either the mild compression diabetic socks or a standard diabetic sock. They will return for four weekly follow up visits.

Additionally a sub-set of 30 subjects will be monitored for changes in physical activity pre and post sock usage. Physical activity monitors will be used to assess daily physical activity for 48hrs prior to receiving the socks and after wearing the socks for four weeks an additional 48hrs will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with lower extremity edema aged 18 or older with the ability and willingness to provide Informed consent
* Patient's ankle-brachial systolic pressure index > 0.6 and toe-brachial index > 0.3
* Patient is willing to participate in all procedures and follow up evaluations necessary to complete the study.
* Patient has diabetes type 1 or type 2 confirmed by patient's primary care physician.

Exclusion Criteria:

* Patients with active wound infection, or untreated osteomyelitis, gangrene
* Patients with dementia, or impaired cognitive function that would prohibit study compliance
* Patients with wide spread malignancy or systemically immuno-compromising disease
* Patients who are unable or unwilling to participate in all procedures and follow up evaluations
* Patient with deep and/or large ulcers that require copious bandaging and may affect efficacy of socks. Patients with superficial ulcers that only require a light dressing are not excluded. The ulcer, if present, must be superficial and cannot exhibit any clinical signs of infection
* Patients with restless leg syndrome, Parkinson's disease, or other disease that will cause involuntary movement during microvascular assessment
* Patients with severe edema or calf circumference greater than 24" or 46cm
* Patients with severe lymphedema
* Patients with edema that in the opinion of the investigator requires higher compression than the 18-25mmHg provided by the compression socks
* Patients who are currently wearing compression hose. (Patients who have been prescribed compression hose but have not worn compression stockings for the past 6 months can be included in the study)
* Patients unable to walk one hundred feet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Wu, DPM, MS, Principal Investigator — Rosalind Franklin University of Medicine and Science
Locations (1):
- Rosalind Franklin University Health System, North Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mild Compression Diabetic Sock | Standard Diabetic Sock
Started | 40 | 40
Received Intervention | 39 (1 participant failed to show up to treatment allocation visit and was subsequently lost to follow up) | 40
Completed | 38 | 39
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mild Compression Diabetic Sock | Standard Diabetic Sock | Total
Number analyzed (Participants) | 38 | 39 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (13) | 64 (13) | 64 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 37
  Male | 20 | 20 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 10 | 25
  White | 19 | 26 | 45
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 38 | 39 | 77
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 34.3 (6.3) | 35.6 (7.4) | 35.0 (6.9)

OUTCOME MEASURES:

1. Primary Outcome: Cutaneous Water Content
Description: Cutaneous water content was measured non-invasively by tissue dielectric constant (MoistureMeter) at a single location: 2 inches distal and 2 inches lateral to the fibular head.
Time Frame: change from baseline after 4 weeks of sock usage
Measure: Mean (95% Confidence Interval); unit: percentage change in dielectric constant
Arm/Group | Mild Compression Diabetic Sock | Standard Diabetic Sock
Number analyzed (Participants) | 38 | 39
percentage change in dielectric constant
  change after 1 week | -1.1 [-3.4 to 1.2] | -.82 [-2.9 to 1.2]
  change after 2 weeks | -0.99 [-3.2 to 1.2] | -2.1 [-4.6 to 0.4]
  change after 3 weeks | -0.23 [-2.4 to 2.0] | -1.7 [-4.0 to 0.57]
  change after 4 weeks | -.16 [-2.2 to 1.8] | -1.6 [-3.7 to 0.46]
Statistical Analysis 1: Comparison: Mild Compression Diabetic Sock vs Standard Diabetic Sock; Test type: Superiority or Other; p > 0.05, ANOVA — 0.05 set as a priori threshold for statistical significance; Sidak correction for multiple comparisons used

2. Primary Outcome: Calf Edema
Description: The circumference of calf was measured by a tape measure.
Time Frame: change from baseline after 4 weeks of sock usage
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | Mild Compression Diabetic Sock | Standard Diabetic Sock
Number analyzed (Participants) | 38 | 39
cm
  change after 1 week | -0.48 [-1.2 to 0.20] | -0.73 [-1.7 to 0.24]
  change after 2 weeks | -0.89 [-1.7 to -0.09] | -0.82 [-1.9 to 0.21]
  change after 3 weeks | -0.75 [-1.6 to 0.14] | -0.85 [-1.9 to 0.2]
  change after 4 weeks | -0.95 [-1.8 to -.07] | -.74 [-1.8 to 0.30]
Statistical Analysis 1: Comparison: Mild Compression Diabetic Sock vs Standard Diabetic Sock; Test type: Superiority or Other; p < 0.05, ANOVA — 0.05 set as a priori threshold for statistical significance; Sidak correction for multiple comparisons used

3. Primary Outcome: Ankle Edema
Description: The circumference of ankle was measured by a tape measure.
Time Frame: change from baseline after 4 weeks of sock usage
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | Mild Compression Diabetic Sock | Standard Diabetic Sock
Number analyzed (Participants) | 38 | 39
cm
  change after 1 week | -0.42 [-1.02 to 0.19] | -0.15 [-0.57 to 0.27]
  change after 2 weeks | -0.68 [-1.1 to -0.22] | -0.28 [-0.80 to 0.24]
  change after 3 weeks | -0.85 [-1.4 to -0.31] | -0.30 [-0.87 to 0.27]
  change after 4 weeks | -.78 [-1.4 to -.019] | -0.34 [-1.0 to 0.36]
Statistical Analysis 1: Comparison: Mild Compression Diabetic Sock vs Standard Diabetic Sock; Test type: Superiority or Other; p < .05, ANOVA — 0.05 set as a priori threshold for statistical significance; Sidak correction for multiple comparisons used

4. Primary Outcome: Toe Brachial Index
Description: ratio of systolic blood pressure of toe relative to systolic blood pressure of arm
Time Frame: change from baseline after 4 weeks of sock usage
Measure: Mean (95% Confidence Interval); unit: unit-less ratio data
Arm/Group | Mild Compression Diabetic Sock | Standard Diabetic Sock
Number analyzed (Participants) | 38 | 39
unit-less ratio data
  change after 1 week | -0.02 [-0.2 to 0.06] | 0.05 [-0.03 to 0.12]
  change after 2 weeks | 0.00 [-0.06 to 0.06] | 0.07 [0.008 to 0.14]
  change after 3 weeks | -0.01 [-0.09 to 0.08] | 0.05 [-0.03 to 0.13]
  change after 4 weeks | -0.003 [-0.08 to 0.07] | 0.06 [-0.01 to 0.13]
Statistical Analysis 1: Comparison: Mild Compression Diabetic Sock vs Standard Diabetic Sock; Test type: Superiority or Other; p > 0.05, ANOVA — 0.05 set as a priori threshold for statistical significance; Sidak correction for multiple comparisons used

5. Primary Outcome: Ankle Brachial Index
Description: ratio of systolic blood pressure of ankle relative to systolic blood pressure of arm
Time Frame: change from baseline after 4 weeks of sock usage
Measure: Mean (95% Confidence Interval); unit: unit-less ratio data
Arm/Group | Mild Compression Diabetic Sock | Standard Diabetic Sock
Number analyzed (Participants) | 38 | 39
unit-less ratio data
  change after 1 week | 0.01 [-0.04 to 0.06] | 0.03 [-0.02 to 0.08]
  change after 2 weeks | 0.01 [-0.05 to 0.07] | 0.05 [-0.01 to 0.1]
  change after 3 weeks | -0.01 [-0.07 to 0.05] | 0.03 [-0.01 to 0.08]
  change after 4 weeks | 0.01 [-0.06 to 0.07] | 0.01 [-0.05 to 0.07]
Statistical Analysis 1: Comparison: Mild Compression Diabetic Sock vs Standard Diabetic Sock; Test type: Superiority or Other; p > 0.05, ANOVA — 0.05 set as a priori threshold for statistical significance; Sidak correction for multiple comparisons used

6. Primary Outcome: Foot Edema
Description: The circumference of the foot was measured by a tape measure.
Time Frame: change from baseline after 4 weeks of sock usage
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | Mild Compression Diabetic Sock | Standard Diabetic Sock
Number analyzed (Participants) | 38 | 39
cm
  change after 1 week | -0.1 [-0.6 to 0.3] | -0.003 [-1.02 to 1.01]
  change after 2 weeks | -0.1 [-0.5 to 0.4] | -0.19 [-1.17 to 0.79]
  change after 3 weeks | -0.2 [-0.7 to 0.3] | -0.36 [-1.5 to 0.75]
  change after 4 weeks | -0.4 [-0.9 to 0.1] | -0.24 [-1.3 to 0.85]
Statistical Analysis 1: Comparison: Mild Compression Diabetic Sock vs Standard Diabetic Sock; Test type: Superiority or Other; p > 0.05, ANOVA — 0.05 set as a priori threshold for statistical significance; Sidak correction for multiple comparisons used

7. Secondary Outcome: Physical Activity Level
Description: Physical activity monitors will be used to assess physical activity patters of participants for 48 hours prior to initiating sock usage and for 48 hours after the participants have worn the socks for four weeks.
Time Frame: baseline and after four weeks of wearing the socks
Population: physical activity measurements were only made for a sub-sample of the study's complete sample
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | Mild Compression Diabetic Sock | Standard Diabetic Sock
Number analyzed (Participants) | 13 | 14
steps
  48hr step count at baseline | 16781.8 (14474.6) | 16984.9 (8559.8)
  48hr step count after 4 weeks | 18056.5 (7360.9) | 15701.0 (6749.7)

8. Primary Outcome: Microcirculation for Medial Calf
Description: microcirculation as measured by skin perfusion pressure
Time Frame: change from baseline after 4 weeks of sock usage
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Mild Compression Diabetic Sock | Standard Diabetic Sock
Number analyzed (Participants) | 38 | 39
mmHg
  change after 1 week | 5.9 [-1.2 to 13.0] | 1.9 [-5.3 to 9.0]
  change after 2 weeks | 7.3 [-0.2 to 14.8] | 3.6 [-5.7 to 12.9]
  change after 3 weeks | 6.5 [-1.3 to 14.4] | -0.71 [-7.4 to 6.0]
  change after 4 weeks | 4.8 [-3.1 to 12.8] | 2.3 [-7.1 to 11.8]
Statistical Analysis 1: Comparison: Mild Compression Diabetic Sock vs Standard Diabetic Sock; Test type: Superiority or Other; p > 0.05, ANOVA — 0.05 set as a priori threshold for statistical significance; Sidak correction for multiple comparisons used

9. Primary Outcome: Microcirculation for Lateral Calf
Description: microcirculation as measured by skin perfusion pressure
Time Frame: change from baseline after 4 weeks of sock usage
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Mild Compression Diabetic Sock | Standard Diabetic Sock
Number analyzed (Participants) | 38 | 39
mmHg
  change after 1 week | 4.4 [-1.9 to 10.8] | 2.6 [-1.5 to 6.7]
  change after 2 weeks | 4.8 [-5.7 to 15.3] | 3.5 [-0.36 to 7.4]
  change after 3 weeks | 7.4 [-2.4 to 17.3] | 0.23 [-4.5 to 5.0]
  change after 4 weeks | 4.4 [-5.7 to 14.4] | -1.1 [-6.3 to 4.0]
Statistical Analysis 1: Comparison: Mild Compression Diabetic Sock vs Standard Diabetic Sock; Test type: Superiority or Other; p > 0.05, ANOVA — 0.05 set as a priori threshold for statistical significance; Sidak correction for multiple comparisons used

10. Primary Outcome: Microcirculation for Dorsum of Foot
Description: microcirculation as measured by skin perfusion pressure
Time Frame: change from baseline after 4 weeks of sock usage
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Mild Compression Diabetic Sock | Standard Diabetic Sock
Number analyzed (Participants) | 38 | 39
mmHg
  change after 1 week | -1.7 [-8.4 to 5.0] | 1.8 [-5.5 to 9.0]
  change after 2 weeks | 3.4 [-4.0 to 10.7] | 0.26 [-7.0 to 7.6]
  change after 3 weeks | 2.6 [-6.4 to 11.6] | 0.03 [-8.1 to 8.2]
  change after 4 weeks | 0.13 [-7.5 to 7.8] | 3.9 [-4.2 to 11.9]
Statistical Analysis 1: Comparison: Mild Compression Diabetic Sock vs Standard Diabetic Sock; Test type: Superiority or Other; p > 0.05, ANOVA — 0.05 set as a priori threshold for statistical significance; Sidak correction for multiple comparisons used

ADVERSE EVENTS:
Arm/Group | Mild Compression Diabetic Sock | Standard Diabetic Sock
Serious Adverse Events (participants affected / at risk) | 2/38 | 1/39
Other Adverse Events (participants affected / at risk) | 4/38 | 6/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mild Compression Diabetic Sock (N=38) | Standard Diabetic Sock (N=39)
spine infection C2-C5 (Infections and infestations) | 1 (1) | 0 (0)
excessive fluid retention (Vascular disorders) | 1 (1) | 0 (0)
fluid retention and hypertension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mild Compression Diabetic Sock (N=38) | Standard Diabetic Sock (N=39)
blister on toe (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
fall induced knee pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
lower extremity numbness (Nervous system disorders) | 0 (0) | 1 (1)
cold (General disorders) | 0 (0) | 1 (1)
shingles (Infections and infestations) | 0 (0) | 1 (1)
pruritic lesions (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
cramping in feet (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
skin irritation (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
cramping in calf (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No